CLINICAL TRIAL: NCT03413423
Title: Secondary Prevention Following Acute Coronary Syndrome Using Integrated Smoking Cessation and Mood Management
Brief Title: Post Acute Cardiac Event Smoking (PACES) Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Minneapolis Heart Institute Foundation (Other); The Miriam Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Minnesota (Other)
Responsible Party: Principal Investigator, Andrew Busch, Senior Investigator, Hennepin Healthcare Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-4375; 1R01HL136327 (NIH)
Record Dates: First submitted 2018-01-19; First posted 2018-01-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndrome; Tobacco Use
Keywords: smoking; depression; Behavioral Activation; Mood management; Secondary Prevention
MeSH Terms: conditions — Acute Coronary Syndrome; Tobacco Use; Smoking; Depression | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAT-CS (Experimental): Participants will receive standard smoking cessation plus Behavioral Activation based mood management. Will be offered the nicotine patch if medically cleared.
  Interventions: Behavioral: BAT-CS
- Smoking Cessation and Health & Wellness (Active Comparator): Participants will receive standard smoking cessation plus health and wellness education. Will be offered the nicotine patch if medically cleared.
  Interventions: Behavioral: Smoking Cessation and Health & Wellness

INTERVENTIONS:
Behavioral: BAT-CS — All participants will receive one hour standard smoking cessation counseling during their hospitalization for an acute coronary syndrome. Participants will be randomized 1 week after discharge. Those assigned to BAT-CS condition will receive 5 more counseling sessions over the 12 weeks after discharge. The first will be up to one hour and will be conducted in person. The next 4 sessions will occur by phone and will take about 30 minutes. Post-discharge sessions will be focused on smoking cessation and mood management using behavioral activation techniques. Participants will be offered the nicotine patch if medically cleared.
  Other Names: Smoking Cessation and Mood Management
  Arms: BAT-CS
Behavioral: Smoking Cessation and Health & Wellness — All participants will receive one hour of standard smoking cessation counseling during their hospitalization for an acute coronary syndrome. Participants will be randomized 1 week after discharge. Those assigned to the Smoking Cessation plus Health and Wellness condition will receive 5 more counseling sessions over the 12 weeks after hospital discharge. The first will be up to one hour and will be conducted in person. The next 4 sessions will occur over the phone and will take about 30 minutes. Post-discharge sessions will be focused on smoking cessation and didactic health and wellness education. Participants will be offered the nicotine patch if medically cleared.
  Arms: Smoking Cessation and Health & Wellness

SUMMARY:
Summary of the Project :

Quitting smoking following acute coronary syndrome (ACS) can reduce mortality up to 50%. However, depression and smoking are highly co-morbid and depressed mood may interfere with cessation and independently predicts mortality. Thus, a single, integrated treatment for both smoking and depression could be highly effective in reducing post-acute coronary syndrome mortality. Behavioral Activation (BA) is a well established treatment for depression and has recently shown promise as a treatment for smoking cessation. The investigators systematically developed an intervention integrating gold standard smoking cessation counseling with existing BA based mood management techniques for post-ACS smokers; Behavioral Activation Treatment for Cardiac Smokers (BAT-CS).

Objective: For this R01 the investigators will evaluate the efficacy of using a single, integrated treatment that targets both depressed mood and smoking (BAT-CS).

DETAILED DESCRIPTION:
This project will implement a fully powered efficacy trial enrolling 324 smokers with ACS and randomize them to 12 weeks of either Behavioral Activation Treatment for Cardiac Smokers (BAT-CS) or control condition (including contact match). BAT-CS interventions will focus on smoking cessation and mood management, while the control condition will focus on smoking cessation and general health education. Both groups will be offered the nicotine patch if medically safe. Follow-up assessments will be conducted at end-of-treatment (12 weeks post-discharge for index event), and 6, 9, and 12 months after hospital discharge. The occurrence of major adverse cardiac events and all-cause mortality will be tracked for up to 60 months post discharge.

ELIGIBILITY:
Inclusion Criteria:

* hospital inpatients with an ACS diagnosis documented in medical record within the past 30 days
* smoked equal or greater than 1 cigarette per day before being hospitalized
* age of 18-75 years
* English fluency
* willing to consider quitting smoking at discharge
* has a telephone or is willing to use a study issued cell phone
* willing to consent to all study procedures.

Exclusion Criteria:

* limited mental competency
* presence of severe mental illness that would interfere with participation or suicidality
* expected discharge to hospice or greater than 50% chance of 6 month mortality per risk calculator
* currently attending counseling for depression or smoking cessation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence abstinence from smoking | 12 Months
  Self-report of no smoking, not even a puff, for 7 days; then Bio-chemically confirmed with saliva cotinine or by carbon monoxide in a breath sample
Depression Symptoms | 12 Months
  The 9 item Patient Health Questionnaire (PHQ-9) ranges from 0-27 with higher scores indicating higher depression symptoms.

SECONDARY OUTCOMES:
Continuous Abstinence From Smoking Since Hospital Discharge | 12 Months
  No smoking, not even a puff, since hospital discharge
Time to Smoking Relapse | 12 Months
  Time in days to first relapse (i.e., smoking on 7 consecutive days or smoking in 2 consecutive 7 day periods), which were determined through timeline follow back interviewing.
Time to Smoking Lapse | 12 Months
  Time in days to first lapse (i.e., first puff of a cigarette) after discharge, which were determined through timeline follow back interviewing.
Depressed mood | The 10 item Center for Epidemiologic Studies Depression Scale ranges from 0-30 with higher scores indicating higher depression symptoms.
  10 Item Center for Epidemiologic Studies Depression Scale (CESD)
Positive Affect | 12 Months
  As measured by the 10 item Positive Affect Negative Affect Scales (PANAS). The positive affect scale on the PANAS ranges from 5-25 with higher scores indicating greater positive affect.
Negative Affect | 12 Months
  As measured by the 10 item Positive Affect Negative Affect Scales (PANAS). The negative affect scale on the PANAS ranges from 5-25 with higher scores indicating greater negative affect.
Systolic and Diastolic Blood Pressure | 12 Months
  Resting Systolic and Diastolic Blood Pressure
Blood Bio-markers | 12 Months
  HDL, LDL, High Sensitivity C-reactive protein, and Fibrinogen
Major adverse cardiac events (MACE) and all cause mortality | 5 years
  Time in days to MACE or all cause mortality. MACE = non-fatal myocardial infarction (using standard American Heart Association definitions), hospitalization for unstable angina, or urgent coronary revascularization.
Health Related Quality of Life | 12 Months
  12-Item Short Form Health Survey (SF-12)
Treatment Acceptability | 12 weeks
  Client Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Busch, PhD, Principal Investigator — Senior Investigator
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Completely de-identified data (i.e.,data that has been cleaned of all 18 types of HIPAA identifiers) will be available to other qualified researchers. Within 18 months of study completion, we will make datasets available to interested investigators who submit a written request to the PI. The only contingency on the use of the data will be that ethical guidelines be followed (e.g., only individuals who have completed a research ethics training course will have access to the data, the data will be stored securely). The NIH will be notified of transmissions of the data to interested investigators.

REFERENCES:
- [Background] Adkins-Hempel M, Japuntich SJ, Chrastek M, Dunsiger S, Breault CE, Ayenew W, Everson-Rose SA, Nijjar PS, Bock BC, Wu WC, Miedema MD, Carlson BM, Busch AM. Integrated smoking cessation and mood management following acute coronary syndrome: Protocol for the post-acute cardiac event smoking (PACES) trial. Addict Sci Clin Pract. 2023 May 12;18(1):29. doi: 10.1186/s13722-023-00388-9. PMID 37173792
- See also: Protocol paper — https://ascpjournal.biomedcentral.com/articles/10.1186/s13722-023-00388-9